CLINICAL TRIAL: NCT05077358
Title: Intracorporeal Versus Extracorporeal Anastomosis In Laparoscopic Right Colon Resection: A Prospective Randomized Multi-center Clinical Trial
Brief Title: Intracorporeal Versus Extracorporeal Anastomosis In Laparoscopic Right Colon Resection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2020-1037
Record Dates: First submitted 2021-08-23; First posted 2021-10-14 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-09

CONDITIONS: Adenocarcinoma of the Colon
Keywords: Intracorporeal anastomosis; Laparoscopic colectomy; Complete mesocolic excision with central vessel ligation; Surgical site infection
MeSH Terms: conditions — Colonic Neoplasms; Surgical Wound Infection

STUDY DESIGN:
Intervention Model Description: This study is a prospective, randomized, multi-center study comparing intracorporeal versus extracorporeal anastomosis in performing laparoscopic right colectomy. The study subjects will be randomly assigned to: 1. Intracorporeal anastomosis 2. Extracorporeal anastomosis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intracorporeal anastomosis (Experimental): In this group, the anastomosis is performed inside the abdominal cavity with a laparoscopic technique. Specimen extraction will be done through Pfannenstiel incision or similar incision in lower abdomen.
  Interventions: Procedure: Intracorporeal anastomosis
- Extracorporeal anastomosis (Active Comparator): In this group, the anastomosis is performed by pulling out the bowel through a laparotomy.
  Interventions: Procedure: Extracorporeal anastomosis

INTERVENTIONS:
Procedure: Intracorporeal anastomosis — In this group, the anastomosis is performed inside the abdominal cavity with a laparoscopic technique. Specimen extraction will be done through Pfannenstiel incision or similar incision in lower abdomen.
  Arms: Intracorporeal anastomosis
Procedure: Extracorporeal anastomosis — In this group, the anastomosis is performed by pulling out the bowel through a laparotomy.
  Arms: Extracorporeal anastomosis

SUMMARY:
STUDY DESIGN This study is a prospective, randomized, multi-center study comparing intracorporeal versus extracorporeal anastomosis in performing laparoscopic right colectomy. The study subjects will be randomly assigned to 1. intracorporeal anastomosis (experimental group) 2. extracorporeal anastomosis (control group) with 1:1 manner. After surgery the subjects will be followed up at 1month, after then, every 3 month in total 3 years.

STUDY POPULATION

1. Screening A detailed review of the medical records will be performed to assess inclusion/exclusion criteria for all subjects who have been diagnosed with right colon tumor (malignant or benign) or benign disease (complicated diverticulitis and so on) that are subject to a right colectomy procedure.

All patients who are eligible, meet the inclusion and none of the exclusion criteria of this study, will be offered enrollment into the study at each site.

RISK ANALYSIS

1. Potential risks All these procedures are in practice today and only surgeons competent in a technique shall be allowed to perform those surgeries. Therefore, there are no anticipated additional risks than would normally be encountered from these surgeries when they are performed for these patients.
2. Potential benefits There may be some benefit due to having closer follow-up in the study.

QUALIFICATION OF PARTICIPATING SURGEONS

1. Surgical procedure

   * Laparoscopic surgery: a surgical technique where operations are performed far from their target anatomy location through small incisions normally less than 15mm.
   * Extracorporeal anastomosis: the anastomosis is performed by pulling out the bowel through a laparotomy.
   * Intracorporeal anastomosis: the anastomosis is performed inside the abdominal cavity with a laparoscopic technique. Specimen extraction will be done through Pfannenstiel incision or similar incision in lower abdomen.
2. Procedure standardization and qualification procedure Participating surgeons should complete the learning curve of the procedure and experience at least 50 laparoscopic right colectomy. They are required to be evaluated by the quality control (QC) committee. They should submit their unedited videos of laparoscopic right colectomy and must be accepted by 2 or more of total 3 QC committee members.

STATISTICAL ANALYSIS Based on attaining a success rate of 85% for the primary endpoint, a total of 106 subjects will be required for each group. Accounting for a 5% loss, a total of 241 subjects will be recruited for this study.

DETAILED DESCRIPTION:
STUDY METHODS

1. Ethical committee approval The study protocol, patient informed consent form and other required study documentation will be reviewed and approved by an institutional review board or any other authority body, prior to study start-up.
2. Study duration and enrollment The total study duration will be approximately 5 years. Study enrollment will take approximately 24 months. The study subjects will have a short-term follow-up at 30 and 3 months post procedure, with long term follow-up upto 3 years after surgery. Surveillance will be performed according to standard follow-up guideline after colorectal cancer surgery.
3. Randomization All the enrolled subject will be randomly assigned to one of the study group (intracorporeal or extracorporeal). The randomization will be performed upon the enrollment at the central institution stratifying center on 1:1 manner by a coordinator who is not aware of any clinical information
4. Data collection Data will be collected at baseline, operative procedure, discharge, 1 month, 3 months and 1 year. A screening log will be maintained at each site during the enrollment period, in which all patients eligible for the trial shall be identified. This will be maintained to ensure no patient selection bias occurs within a center or by a surgeon.
5. Informed Consent Using the study-specific, IRB approved, informed consent form, information pertinent to this study will be provided to the subjects in writing and in their native, non-technical, language. The consent form will include a description of the study and its purpose, potential benefits, potential risks, site contact information, and all other elements required of an informed consent.

   Subjects are required to voluntarily sign the informed consent form before any study-specific procedure is performed. The Investigator and/or his/her authorized designee, trained on the protocol and performing a consent, will conduct the informed consent process and will answer questions the subjects may have. If the subject agrees to participate, the informed consent form must be signed and dated by the subject or his/her legally authorized representative prior to enrollment in the study and separately signed and dated by the person taking consent. Only subjects who have signed the study informed consent will be included in the study.
6. Withdrawal and discontinuation The subject's participation in any clinical trial is voluntary. The subject has the right to withdraw at any time without penalty or loss of benefit. Study withdrawal means the subject is no longer participating in the study and no further follow-ups will be performed. All subjects that withdraw after informed consent is signed will be evaluated at the time of withdrawal. Every effort will be made to document the subject outcome at the time of withdrawal. The investigator has the right to discontinue subjects from the study at their discretion to ensure wellbeing of the subject. The reasons for withdrawal shall be documented.

ELIGIBILITY:
Inclusion Criteria:

1. 19 years or older
2. Right colon tumor with indication for right colectomy (malignant disease).
3. Patients with adequate performance status (Eastern Cooperative Oncology Group Scale score of ≤2)
4. Patient has signed and dated the Informed consent before patient inclusion in the study.

Exclusion Criteria:

1. Patient with a comorbid illness or condition that would preclude the use of surgery.
2. Patients with cT4b tumors.
3. Patients whose disease condition requires major simultaneous combined resection other than right colectomy (e.g. other intestinal resection, liver resection)
4. Patients unwilling to comply with all follow-up study requirements
5. Patient undergoing emergency procedures
6. Obstructive disease (but, possible to enroll after stent insertion resolving obstruction)
7. Impossible preoperative bowel preparation
8. Metastatic disease
9. Pregnant or suspected pregnancy
10. Complicated inflammatory bowel disease (Crohn´s Disease, Ulcerative Colitis, Intestinal tuberculosis, Behcet's disease, Undetermined inflammatory bowel disease) that combined with intraabdominal abscess or intestinal fistula
11. No Informed consent

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Estimated)
Dates: Start 2021-04-05 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
surgical site infection | within 30 postoperative days
  The efficacy of the anastomosis technique is defined as a lack of surgical site infection within 30 postoperative days.
  1. Superficial surgical site infection
  2. Deep surgical site infection

SECONDARY OUTCOMES:
3 year disease-free survival | 3 years
Tissue morphometry | within 30 postoperative days
  1. The distance from the tumour and the closest bowel wall to the high vascular tie (mm)
  2. The length of colon and ileum (mm)
  3. The area of mesocolon (mm2)
  4. Macroscopic quality of specimen (3 grades) G1 : intact mesocolon G2 : significant mesocolic disruptions away from the muscularis G3 : significant disruptions extending down to the muscularis
Incidence of incisional hernia within 1 year after surgery | 1 year
Postoperative pain score in visual analogue scale | within 7 postoperative days
Length of postoperative hospital stay | within 7 postoperative days
Number of patient with Clavien-Dindo grade IIIb-IV at 30 days postop as an operation-related morbidity | within 30 postoperative days
Operative time (min) | within the day of operation
Incidence of conversion | within 30 postoperative days

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hellan M, Anderson C, Pigazzi A. Extracorporeal versus intracorporeal anastomosis for laparoscopic right hemicolectomy. JSLS. 2009 Jul-Sep;13(3):312-7. PMID 19793468
- [Background] van Oostendorp S, Elfrink A, Borstlap W, Schoonmade L, Sietses C, Meijerink J, Tuynman J. Intracorporeal versus extracorporeal anastomosis in right hemicolectomy: a systematic review and meta-analysis. Surg Endosc. 2017 Jan;31(1):64-77. doi: 10.1007/s00464-016-4982-y. Epub 2016 Jun 10. PMID 27287905
- [Background] Shapiro R, Keler U, Segev L, Sarna S, Hatib K, Hazzan D. Laparoscopic right hemicolectomy with intracorporeal anastomosis: short- and long-term benefits in comparison with extracorporeal anastomosis. Surg Endosc. 2016 Sep;30(9):3823-9. doi: 10.1007/s00464-015-4684-x. Epub 2015 Dec 10. PMID 26659237
- [Background] Wu Q, Jin C, Hu T, Wei M, Wang Z. Intracorporeal Versus Extracorporeal Anastomosis in Laparoscopic Right Colectomy: A Systematic Review and Meta-Analysis. J Laparoendosc Adv Surg Tech A. 2017 Apr;27(4):348-357. doi: 10.1089/lap.2016.0485. Epub 2016 Oct 21. PMID 27768552
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] Xu H, Li J, Sun Y, Li Z, Zhen Y, Wang B, Xu Z. Robotic versus laparoscopic right colectomy: a meta-analysis. World J Surg Oncol. 2014 Aug 28;12:274. doi: 10.1186/1477-7819-12-274. PMID 25169141